CLINICAL TRIAL: NCT04479943
Title: Preventing Hospital-Acquired Disability: An Intervention to Improve Older Adult Patient Ambulation
Brief Title: Improving Patient Walking During Hospitalization
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-0010; A549000 (Other: UW Madison); NUR/FACULTY AFFAIRS/ADMIN (Other: UW Madison); Protocol Version 08/19/2024 (Other: UW Madison); 1R01HS026733-01A1 (AHRQ)
Record Dates: First submitted 2020-07-14; First posted 2020-07-21 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Early Mobility; Older Adults; Hospital Acquired Condition
Keywords: nursing care; hospitalization; aged; walking
MeSH Terms: conditions — Iatrogenic Disease | interventions — Surveys and Questionnaires; Focus Groups

STUDY DESIGN:
Intervention Model Description: This study uses an incomplete stepped wedge cluster randomized controlled trial. In the incomplete stepped wedge design, inpatient units are randomly sequenced into the intervention. A baseline (control period) and 2 follow up data collection periods (intervention and post intervention period) occur for each unit. Incomplete stepped wedge cluster randomized trials are novel study designs that are particularly beneficial for evaluating service delivery interventions using a pragmatic design, when evaluations need to be completed at a system or population level, or it is impractical or cost prohibitive to roll out an intervention across multiple units simultaneously.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-intervention/control (No Intervention): 160-200 older adult patients (age 65 or older) will be recruited on four units across two hospitals (two units per hospital) over 6-8 months prior to implementation of the unit-based MOVIN intervention.
- Post-intervention (Experimental): 160-200 older adult patients (age 65 or older) will be recruited on four units across two hospitals (two units per hospital) over 6-8 months after MOVIN has been implemented on the unit.
  Interventions: Other: MOVIN
- Nurses (Experimental): Nurses will complete surveys and provide qualitative data to assess barriers to implementation
  Interventions: Other: Surveys and Focus groups

INTERVENTIONS:
Other: MOVIN — MOVIN is a multi-component unit-based intervention comprised of five components that are implemented simultaneously in a hospital unit. The five components are: 1) psychomotor skills training, 2) unit ambulation culture, 3) communication, 4) resources, 5) ambulation environment.
  Arms: Post-intervention
Other: Surveys and Focus groups — Nurses will answer surveys about nurse behavior, changes in self-efficacy, frequency and distance of patient ambulation, documentation of ambulation, qualitative data collected to determine barriers to implementation
  Arms: Nurses

SUMMARY:
The MOVIN (Mobilizing Older adult patients Via a systems-based Intervention) randomized controlled trial is designed to evaluate the impact of the MOVIN intervention on improving the functional ability of older adult hospital patients and reducing their healthcare utilization post-hospitalization. MOVIN is a program to increase patient ambulation while hospitalized. The study's hypothesis is that MOVIN will improve functional outcomes for hospitalized older adult patients by producing a change in nursing practice and culture of ambulation on inpatient units. MOVIN is a unit-based intervention. Therefore all patients on this unit are exposed to the intervention once it is implemented regardless of whether or not they participate in the trial. The study will enroll 360-420 total hospitalized participants 65 years and older for the duration of their stay.

DETAILED DESCRIPTION:
Up to 65% of hospitalized older adults will lose the ability to ambulate independently during their hospital stay. Loss of independent ambulation has been identified as a hospital-acquired disability and is a critical patient safety concern, resulting in permanent loss of function for 50% of older adults one-year post discharge. Functional loss is associated with multiple negative outcomes including a 33% increase in new nursing home placement, increase in length of hospital stay, need for home health services, falls, caregiver burden, decreased quality of life, and increased mortality. Given the rapid increase in the elderly population, loss of independent ambulation primarily due to the process of care in hospital settings may significantly increase future healthcare costs and further exacerbate concerns related to patient care quality.

Lack of walking during hospitalization has been directly linked to loss of independent ambulation in older adults. Nurses are responsible for promoting and maintaining patient independent mobility. However, the investigators research has identified multiple personal and organizational barriers that prevent nurses from walking patients. The investigators have developed and pilot tested a novel systems based multi-component intervention to improve ambulation of older adult patients, Mobilizing Older adult patients Via a systems-based INtervention (MOVIN).

MOVIN is comprised of five components: 1) psychomotor skills training; 2) communication tools; 3) ambulation pathways; 4) ambulation resources; and 5) unit ambulation culture. The Investigators pilot study of MOVIN demonstrated a statistically significant increase in frequency and weekly distance of patient ambulation as well as changes in nursing practice and unit culture. Notably, these changes have been sustained for greater than two years after completion of the study.

The investigators' goal is to eliminate loss of independent ambulation in hospitalized older adults. In pursuit of this goal, the specific aims are to:

* Specific Aim 1:Test the effectiveness of MOVIN to improve functional ability of older adult patients at discharge, and 1, 3 and 6 months post discharge
* Specific Aim 2: Test the effectiveness of MOVIN to reduce healthcare utilization of older adults at discharge, and 1, 3 and 6 months post discharge

  * 2.A. To analyze a return on investment of MOVIN based on program costs and health utilization measures across different hospitals
* Specific Aim 3: Measure change in nurse behaviors and unit culture and identify ongoing systems barriers that impact translation of MOVIN across inpatient units and different hospitals.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or older
* able to walk with or without assistance
* living in the community (not long term care) prior to admission
* have an ambulation order
* admitted to hospital's general adult medical unit
* able to consent
* able to speak and understand English
* at least 24h planned length of stay after initial study enrollment.

Exclusion Criteria:

* activated Power of Attorney
* lower extremity amputation
* on hospice
* bed rest order or activity restriction
* wheelchair bound

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 387 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Change in gait speed | Within 24 hours of hospital admission, Within 8 hours of hospital discharge, 1 month post-discharge, 3 months post-discharge; Up to 4 months total
  Gait Speed is a physical performance measure identified as a sensitive clinical indicator of health, mortality, healthcare utilization, and independence in ambulation, and is feasible to test in hospitalized older adults. A 4 meter walk test will be conducted on admission to the study, discharge from the hospital and at 3 months post discharge in the subjects home or the hospital or clinic. A trained member of the research team will conduct the gait speed test. Interrater reliability for the 4 meter walk test will be conducted between all members of the research team prior to collecting gait speed data on study participants. Change scores will be calculated as the difference among gait speeds measured at each time points.
Aim 1: Change in self-report on Activities of Daily Living (ADL) | Within 24 hours of hospital admission, Within 8 hours of hospital discharge, 1 month post-discharge, 3 months post-discharge; 6 months post-discharge; Up to 7 months total
  A trained member of the research team will collect patients self-report of ADLs on admission to the study, discharge from the hospital, by phone at 1 month post intervention and 6 months post intervention, and in person at the 3 month post intervention visit using the Katz ADL Index. The Katz ADL Index is a self-report scale that measures five ADL on three levels (independent, requiring assistance of another and unable to do). A score of 0-6 is possible, with higher scores indicating higher independence with ADLs and lower scores indicating higher dependence on others to perform ADLs. The scale demonstrates excellent reliability and predictive validity, and is sensitive to change in hospital settings. Change scores will be calculated as the difference among ADL independence measured at each time point.
Aim 1: Change in Life Space Assessment | Within 24 hours of hospital admission, Within 8 hours of hospital discharge, 1 month post-discharge, 3 months post-discharge; 6 months post-discharge; Up to 7 months total
  The UAB Life Space Assessment (LSA) is a self-report scale of ambulation that measures spaces patients' move in, the frequency of moving into those spaces, and dependency in moving into those spaces. This scale has demonstrated reliability and predictive validity and sensitivity to change after hospital stay. Level scores are calculated by multiplying the life-space level (higher numbers indicate farther distances moved, e.g., 1-inside the home to 5-places outside of the person's town), degree of independence (higher scores indicate greater independence), and frequency of movement (higher scores equal greater frequency). Total scores range from 0 (totally bed-bound) to 120 (moved out of town every day without assistance). A trained member of the research team will collect patients self-report on Life Space. Change scores will be calculated as the difference among LSA ambulation measured at each time point.
Aim 2: Hospital Readmissions | 1 month post-discharge; 3 months post-discharge; 6 months post-discharge; Up to 7 months total
  Hospital readmissions will be collected via patient self-report and via medical record review by a trained researcher from the study team.
Aim 2: Emergency Room Visits | 1 month post-discharge; 3 months post-discharge; 6 months post-discharge; Up to 7 months total
  Emergency room visits Discharge destination (home, skilled nursing facility) will be collected via patient self report.
Aim 2: Length of Hospital Stay | Within 3 months post-discharge; Up to 4 months total
  Length of hospital stay will be collected via patient medical record review by a nurse researcher from the study team.
Aim 2: Discharge Destination | Within 3 months post-discharge; Up to 4 months total
  Discharge destination (home, skilled nursing facility) will be collected via patient medical record review by a nurse researcher from the study team.
Aim 3: Distance of Patient Ambulation | 6 months pre-intervention, during the 14-week intervention period, and 6 months post-intervention; up to 16 months total
  Unit level data on the distance in feet recorded for ambulation events in the electronic health record.
Aim 3: Barriers to Ambulation Survey | pre-intervention, post-intervention (up to about 20 weeks)
  Data collected from enrolled nursing staff via paper copies or online link before and after the intervention. The Barriers to Patient Ambulation Survey assesses the nurses opinions regarding ambulation of hospitalized patients within the past 2 weeks. It is scored from 0-100 with higher scores indicating increased barriers to ambulation.
Aim 3: Ambulation Culture Survey | pre-intervention, post-intervention (up to about 20 weeks)
  Data collected from enrolled nursing staff via paper copies or online link before and after the intervention. The Ambulation Culture Survey asks for opinions on ambulation culture. It is scored by calculating the percent of positive responses across the sample from 0-100% where higher scores indicate better opinion of ambulation culture.
Aim 3: Qualitative Assessment of Intervention Implementation | post-intervention (approximately 3-5 months after active intervention launch)
  Enrolled nursing staff will be interviewed and interviews will be coded for themes. Themes will be summarized to report by participant count.

SECONDARY OUTCOMES:
Patient Satisfaction: Count of Participants With Satisfaction Responses to Never, Sometimes, Usually, Always Questions on HCAHPS | 6 months pre-intervention, during the 14-week intervention period, and 6 months post-intervention; up to 16 months total
  HCAHPS is a participant self-reported survey that measures patient satisfaction. Reported here are Participant Counts to questions with response options: Never, Sometimes, Usually, Always. Analysis will include shifts of distribution across response options and changes in frequency/percentage of top-box responses ("Always") relative to all responses. Questions include:
  During this hospital stay, how often did nurses treat you with courtesy and respect? how often did nurses listen carefully to you? how often did nurses explain things in a way you could understand? after you pressed the call button, how often did you get help as soon as you wanted it? how often were your room and bathroom kept clean? how often was the area around your room quiet at night? How often did you get help in getting to the bathroom or in using a bedpan as soon as you wanted?
Patient Satisfaction: Count of Participants Answering Yes to items on the HCAPHS | 6 months pre-intervention, during the 14-week intervention period, and 6 months post-intervention; up to 16 months total
  The HCAPHS is a participant self-reported survey that measures patient satisfaction. Reported here are the Participant Counts of those who answered "Yes" to the following Yes or No questions:
  * During this hospital stay, did you need help from nurses or other hospital staff in getting to the bathroom or in using a bedpan?
  * During this hospital stay, were you given any medicine that you had not taken before?
  * During this hospital stay, did doctors, nurses, or other hospital staff talk with you about whether you would have the help you needed when you left the hospital?
  * During this hospital stay, did you get information in writing about what symptoms or health problems to look out for after you left the hospital?
  * During this hospital stay, were you admitted to this hospital through the Emergency Room?
  * Were you visited by a member of our nursing leadership team during your stay?
Patient Satisfaction: Where Participants Went After Hospitalization | 6 months pre-intervention, during the 14-week intervention period, and 6 months post-intervention; up to 16 months total
  The HCAPHS is a participant self-reported survey that measures patient satisfaction. Reported here are the Participant Counts of whether they went home, to someone else's home, or another facility after discharge.
Patient Satisfaction: Hospital Experience Scores from 0-10 on HCAPHS | 6 months pre-intervention, during the 14-week intervention period, and 6 months post-intervention; up to 16 months total
  The HCAPHS is a participant self-reported survey that measures patient satisfaction. Participants rank their hospital experience from 0-10, where 10 is the best possible hospital.
Patient Satisfaction: Count of Participants With Satisfaction Responses to Definitely no/Probably no/Probably yes/Definitely yes to the following question: Would you recommend this hospital to your friends and family? | 6 months pre-intervention, during the 14-week intervention period, and 6 months post-intervention; up to 16 months total
  The HCAHPS is a participant self-reported survey that measures patient satisfaction. Reported here are the Participant Counts With Satisfaction Responses to Definitely no/Probably no/Probably yes/Definitely yes to the following question: Would you recommend this hospital to your friends and family? Analysis will include shifts in the distribution of responses across response options, as well as changes in frequency/percentage of top-box responses (responses of "Definitely Yes") relative to all responses.
Patient Satisfaction: Count of Participants With Responses to Strongly disagree/Disagree/Agree/Strongly agree questions on HCAHPS | 6 months pre-intervention, during the 14-week intervention period, and 6 months post-intervention; up to 16 months total
  The HCAHPS is a participant self-reported survey that measures patient satisfaction. Reported here are the Participant Counts of Responses to Strongly disagree/Disagree/Agree/Strongly agree to the following questions:
  During this hospital stay, staff took my preferences and those of my family or caregiver into account in deciding what my health care needs would be when I left When I left the hospital, I had a good understanding of the things I was responsible for in managing my health When I left the hospital, I clearly understood the purpose for taking each of my medications
  Analysis will include shifts in the distribution of responses across response options, as well as changes in frequency/percentage of top-box responses (responses of "Strongly agree") relative to all responses.
Patient Satisfaction: Participant Experience Scores from 1-5 on HCAHPS | 6 months pre-intervention, during the 14-week intervention period, and 6 months post-intervention; up to 16 months total
  The HCAPHS is a participant self-reported survey that measures patient satisfaction. Participants rank their hospital experience from 1-5, where 5 is the best possible experience.
Aim 2: Physical Therapy (PT) Utilization | 6 months pre-intervention, during the 14-week intervention period, and 6 months post-intervention; up to 16 months total
  Billing data will be used retrospectively to understand use of PT services on the intervention units at pre-intervention, intervention, and post-intervention data collection periods
Aim 3: Frequency of Patient Ambulation (times per day) | 6 months pre-intervention, during the 14-week intervention period, and 6 months post-intervention; up to 16 months total
  Unit-level data on the number of times an ambulation event is recorded by nursing staff in the electronic health record.
Aim 3: Nurse Fatigue Survey | pre-intervention, post-intervention (up to about 20 weeks)
  Data collected from enrolled nursing staff via paper copies or online link before and after the intervention. The Nurse Fatigue Survey measures experience of fatigue and strain at work and home. It is a 15 item survey scored on a 7 point likert scale from 0 (strongly disagree) to 6 (strongly agree) with the 3 subscales of 5 questions each (chronic fatigue, acute fatigue and intershift recovery) scored separately. Items for each subscale are aggregated into a percent of the total highest possible points (30) resulting in a range of scores from 0-100%, higher scores indicate higher fatigue.
Aim 3: Professional Quality of Life Survey | pre-intervention, post-intervention (up to about 20 weeks)
  Data collected from enrolled nursing staff via paper copies or online link before and after the intervention. The Professional Quality of Life Survey measures positive and negative experiences within the last 30 days in a 30-item survey scored on a 5 point likert scale from 1 (never) to 5 (very often). There are 3 subscales: Compassion Satisfaction, Burnout, and Secondary Traumatic Stress, each subscale has a range of scores from 10-50, with higher scores indicative of higher compassion satisfaction, higher burnout, and higher secondary traumatic stress.

CONTACTS AND LOCATIONS:
Overall Officials: Linsey M Steege, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No